CLINICAL TRIAL: NCT07181135
Title: A Parallel-group, Randomized, Prospective, Interventional, Double-blind, Multicenter Global Phase 3 Study to Investigate the Efficacy and Safety of Finerenone Versus Placebo, in Participants With Chronic Kidney Disease Not Using Renin-angiotensin-system Inhibitors
Brief Title: FINE-START: Efficacy and Safety of Finerenone in Patients With Chronic Kidney Disease Not Using Renin-angiotensin-system Inhibitors
Acronym: FINE-START
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22817; 2025-523075-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-09; First posted 2025-09-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease
Keywords: kidney disease; albuminuria; Finerenone
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Albuminuria | interventions — finerenone

STUDY DESIGN:
Intervention Model Description: parallel-group, randomized, prospective, interventional, double-blind study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone (Experimental): Finerenone 10mg or 20mg, tablet (oral), once daily for approximately 6 months.
  Interventions: Drug: Finerenone (BAY 94-8862)
- Placebo (Placebo Comparator): Placebo matching Finerenone 10mg or 20mg, tablet (oral), once daily for approximately 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY 94-8862) — Finerenone 10 or 20mg in participants with chronic kidney disease not using renin-angiotensin-system inhibitors
  Arms: Finerenone
Drug: Placebo — Placebo matching finerenone
  Arms: Placebo

SUMMARY:
Study to demonstrate efficacy of finerenone when compared to placebo in reducing albuminuria in participants with chronic kidney disease (CKD) not using renin-angiotensin-system (RAS) inhibitors.

DETAILED DESCRIPTION:
FINE-START is a multicenter, international, randomized, placebo-controlled, double blind parallel-group Phase 3 study in adult participants with chronic kidney disease (CKD) not using renin-angiotensin-system (RAS) inhibitors. The study will enroll adults (≥18 years) with CKD defined as eGFR ≥25 and <120 mL/min/1.73 m2, urinary albumin-to-creatinine ratio (UACR) ≥100 mg/g (11.3 mg/mmol) to <5000 mg/g (565 mg/mmol) and documentation of elevated albuminuria or proteinuria. A total of 180 participants will be included and randomized with equal allocation (1:1) to Finerenone or placebo. Finerenone or placebo will be administered once daily for approximately 6 months. Change in UACR from baseline over 6 months will be used as a primary endpoint to demonstrate slowing of kidney disease progression. The aim of this study is to demonstrate efficacy of finerenone when compared to placebo in reducing albuminuria in participants with chronic kidney disease (CKD) not using renin-angiotensin-system (RAS) inhibitors.

ELIGIBILITY:
Main Inclusion Criteria:

1. Adults (≥18 years) with Chronic Kidney Disease defined as:

   * eGFR ≥25 and <120 mL/min/1.73 m2 using CKD-EPI 2009 formula at the Screening visit.
   * UACR ≥100 mg/g (11.3 mg/mmol) to <5000 mg/g (565 mg/mmol) at the Screening visit (geometric mean of the 3 measurements) and documentation of elevated albuminuria or proteinuria.
2. Potassium level ≤5.0 mmol/L at Screening (local assessment).
3. No current or previous (within 8 weeks prior to the Screening visit) treatment with RAS inhibition (ACEi, ARB, or Renin inhibitor (e.g. Aliskiren)).

Main Exclusion Criteria:

1. Participants with an HbA1c>11%.
2. Participants with type 1 diabetes.
3. Symptomatic heart failure with reduced ejection fraction and class 1A indication for MRA treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin-to-creatinine ratio (UACR) | Baseline upto 6 months
  Change in UACR from baseline (ratio to baseline) over 6 months

SECONDARY OUTCOMES:
TEAEs, TESAEs | Baseline upto 6 months
  Number of participants with treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs)
Number of participants with Hyperkalemia | Baseline upto 6 months
  Number of participants with Hyperkalemia (adverse event of special interest, AESI)

CONTACTS AND LOCATIONS:
Overall Officials: Hiddo J. Lambers Heerspink, Prof. Dr., Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: No